CLINICAL TRIAL: NCT00236158
Title: The Danish Multicenter Randomised Study on AAI Versus DDD Pacing in Sick Sinus Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Not able to recruit the estimated number of patients
Sponsor: The DANPACE Investigator Group (Other)
Responsible Party: Henning Rud Andersen, Aarhus University Hospital Skejby, Departm. of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25100; NCT00236158
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Sick Sinus Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AAIR (Other)
  Interventions: Device: AAIR/DDDR pacemaker
- DDDR (Other)
  Interventions: Device: AAIR/DDDR pacemaker

INTERVENTIONS:
Device: AAIR/DDDR pacemaker — Pacemaker with single lead or dual lead

SUMMARY:
Hypothesis Treatment with rate adaptive single chamber atrial pacing (AAIR) reduces the risk of death compared with rate adaptive dual chamber pacing (DDDR) in patients with sick sinus syndrome (SSS).

Primary purpose The primary purpose of this randomised trial is to compare AAIR and DDDR pacing in patients with SSS and normal atrioventricular (AV) conduction with respect to the primary end point overall mortality.

DETAILED DESCRIPTION:
Background In patients with isolated SSS, who need pacemaker treatment, any pacemaker can be used to treat the symptomatic bradycardia: a single chamber atrial (AAI) pacemaker, a single chamber ventricular (VVI) pacemaker, or a dual chamber (DDD) pacemaker. In the USA and in most European countries, DDD pacing is used in most cases. It is now known from the Danish AAI/VVI trial, that AAI pacing is superior to VVI pacing, since VVI pacing is associated with a higher mortality and a higher incidence of atrial fibrillation, thromboembolic complications and heart failure. This confirms previous findings in observational studies. Therefore, VVI pacing should no longer be used in patients with SSS.

The main argument for using DDD pacing is the concern, that the patients will develop symptomatic atrioventricular (AV) block. In the Danish AAI/VVI trial, the risk of AV block was approximately 0.6% per year, which is equivalent to the risk found in a larger meta analysis. This is only a little higher that the risk of atrioventricular block in the age-matched non-paced population. Implantation of a DDD pacemaker in all patients will effectively prevent development of symptomatic bradycardia in the minority of patients who develops AV block. However, the most important disadvantage during DDD pacing is the stimulation (pacing) of the ventricles by the pacemaker a large part of the time, also in patients without AV block. Pacing the right ventricle causes an asynchronous electrical activation and mechanical contraction of the ventricles as compared with the normal physiological contraction.

At present time, a randomised comparison of AAI and DDD pacing in patients with SSS has never been conducted, and to our knowledge, such a trial is not planned anywhere else.

Since several of the patients with SSS suffer from chronotropic incompetence, pacemakers with rate adaptive function are chosen for all patients included in the present trial.

All patients, that fulfils the inclusion criteria and none of the exclusion criteria and who give written informed consent, are included into the study. For all other patients undergoing primary pacemaker implantation in the study period, an exclusion data sheet is filled in stating the reason for exclusion. A total of 1,900 patients are included into the study.

Prior to the pacemaker implantation patients are randomised by lot (envelope) to either AAIR or DDDR pacing. The randomisation is performed after written informed consent has been obtained from the patient. Randomisation will ensure that all centres will randomise an equal number of patients into each treatment group.

Patients randomised to AAIR pacing will have a bipolar lead implanted in their right atrium connected to a single chamber pacemaker with rate adaptive function. Patients randomised to DDDR pacing will have two leads (one bipolar lead in their right atrium and a uni- or bipolar lead in their right ventricle) connected to a DDDR pacemaker.

Out of hospital follow-up The patients must attend for out of hospital follow-up after 3 months and 12 months and then once every year.

Criteria for closing the study

The DANPACE study is stopped and results are analysed when all of the following three criteria are fulfilled:

1. 1,900 patients have been randomised.
2. The last randomised patient has been followed for at least 1 year.
3. The mean follow-up for the whole study population is at least 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

General:

A. Undergoing primary pacemaker implantation B. Able to appear for outpatient follow-up C. Age > 18 years

Symptoms:

D. Syncope or E. Dizzy spells or F. Congestive heart failure

Electrocardiographic:

G. Sinus bradycardia <40/minute for at least 1 minute in a conscious awake state or H. Sinus arrest/sinoatrial block >2 seconds or I. Bradycardia/tachycardia with sinus-pauses >2 seconds

Exclusion Criteria:

Clinical:

A. Malignant disease. B. Severe psychogenic disease including severe decrepitude and dementia. C. Impending larger operation expected to influence the major end point. D. Cardiac disorder expected to need cardiac surgery during the follow-up period.

E. Need for other device implantation: ICD (implantable cardioverter defibrillator) or implantable DC converter (for atrial fibrillation).

F. Carotid sinus syndrome (positive carotid sinus massage with pauses >3 seconds).

Electrocardiographic:

G. Atrioventricular block. H. Bundle-branch block (complete RBBB, LBBB, bifascicular bundle-branch block or non-specific intraventricular block with QRS >0.12 seconds).

I. Chronic atrial fibrillation. J. Atrial fibrillation/atrial flutter with QRS pauses >3 seconds during atrial fibrillation.

K. Atrial fibrillation/atrial flutter with QRS frequency <40/minute for 1 minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 1999-03; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality after a mean follow-up of 5.5 year. | 5,5 years

SECONDARY OUTCOMES:
Cardiovascular death | 5,5 years
Chronic atrial fibrillation | 5,5 years
Paroxysmal atrial fibrillation | 5,5 years
Arterial thromboembolism | 5,5 years
Congestive heart failure | 5,5 years
Need for pacemaker re-operations | 5,5 years
Quality of life | 5,5 years
Health economics | 5,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henning R Andersen, MD, DMSc, Principal Investigator — Skejby Sygehus, Aarhus University Hospital
Locations (1):
- Department of Cardiology, Skejby Sygehus, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Kirkfeldt RE, Andersen HR, Nielsen JC; DANPACE Investigators. System upgrade and its complications in patients with a single lead atrial pacemaker: data from the DANPACE trial. Europace. 2013 Aug;15(8):1166-73. doi: 10.1093/europace/eut039. Epub 2013 Feb 28. PMID 23449923
- [Derived] Nielsen JC, Thomsen PE, Hojberg S, Moller M, Riahi S, Dalsgaard D, Mortensen LS, Nielsen T, Asklund M, Friis EV, Christensen PD, Simonsen EH, Eriksen UH, Jensen GV, Svendsen JH, Toff WD, Healey JS, Andersen HR; DANPACE investigators. Atrial fibrillation in patients with sick sinus syndrome: the association with PQ-interval and percentage of ventricular pacing. Europace. 2012 May;14(5):682-9. doi: 10.1093/europace/eur365. Epub 2011 Nov 20. PMID 22106360
- [Derived] Nielsen JC, Thomsen PE, Hojberg S, Moller M, Vesterlund T, Dalsgaard D, Mortensen LS, Nielsen T, Asklund M, Friis EV, Christensen PD, Simonsen EH, Eriksen UH, Jensen GV, Svendsen JH, Toff WD, Healey JS, Andersen HR; DANPACE Investigators. A comparison of single-lead atrial pacing with dual-chamber pacing in sick sinus syndrome. Eur Heart J. 2011 Mar;32(6):686-96. doi: 10.1093/eurheartj/ehr022. Epub 2011 Feb 7. PMID 21300730